CLINICAL TRIAL: NCT04633733
Title: An Open-label, Multiple-dose, Fixed-sequence, 3-Period Study to Evaluate the Pharmacokinetic Interactions Between HL237 and Tacrolimus in Healthy Male Subjects
Brief Title: The Study of Pharmacokinetic Interactions Between HL237 and Tacrolimus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HL237-103
Record Dates: First submitted 2020-11-13; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: Fixed-sequential
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): This single arm is conducted in fixed-sequence(Treatment A ->(washout period) -> Treatment B -> Treatment C -> Maintenance treatment).
  Treatment A : tacrolimus 5mg po single dose, Treatment B : HL237 400mg bid for 4 days, Treatment C: tacrolimus 5mg po single dose and HL237 400 mg bid, Maintenance treatment : HL237 400mg bid for 2 days
  Interventions: Drug: HL237 tablet; Drug: tacrolimus capsule

INTERVENTIONS:
Drug: HL237 tablet — HL237 400mg will be administered orally twice a day.
Drug: tacrolimus capsule — tacrolimus 5mg will be administered orally once a day.

SUMMARY:
This study aims to evaluate the pharmacokinetic interaction between HL237 and tacrolimus in healthy male subjects.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetic interaction by comparing of pharmacokinetic parameters when administered HL237(or tacrolimus) between with tacrolimus(or HL237) and without tacrolimus(or HL237).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, 19 years ≤ age ≤ 45
* Body weight ≥ 50kg and 18.5 ≤ BMI ≤ 29.9kg/m2
* Subjects are agree to use contraceptives that protocol suggest and not provide sperm for up to 2 months after the last administration of the investigational drug
* Volunteer

Exclusion Criteria:

* Subject with serious cardiovascular, respiratory, hepatology, renal, hematologic, gastrointestinal, immunologic, dermal, neurologic, or psychological disease or history of such disease
* Subject with symptoms of acute disease within 28 days prior to investigational products dosing
* Subject with medical history which able to affect absorption, distribution, metabolism and excretion of drug
* Subject with hypersensitive reaction to following drug or history of clinically significant hypersensitive reaction to following drug

  * Calcineurin inhibitor or Macrolides
  * HL237
* Subject with clinically significant active chronic disease
* Subject with genetic deficiency such as galactose intolerance, Lapp lactose deficiency or glucosegalactose malabsorption
* Subjects who showed one or more of the following in a screening test including a retest

  * AST, ALT > UNL (upper normal limit) x 2.5
  * Creatinine clearance =< 80mL/min (Cockcroft-Gault GFR = (140-age) * (Wt in kg) / (72 * Cr))
  * Results of ECG, QTc > 450 msec
* Positive test results for hepatitis B virus surface antigen, anti-hepatitis C virus antibody, anti-Human Immunodeficiency virus antibody or venereal disease research laboratory test
* Use of any prescription medication within 14 days prior to study medication dosing
* Use of any over-the-counter(OTC) medication within 7 days prior to study medication dosing
* Subject with clinically significant allergic disease (except for mild allergic rhinitis and mild allergic dermatitis that are not needed to administer drug)
* Subject who is not able to taking standard meals provided by the institution
* Subject with whole blood donation within 60 days, component blood donation within 20 days
* Subjects receiving blood transfusion within 30 days prior to study medication dosing
* Participation in any clinical investigation within 6 months prior to study medication dosing
* Use of any medication effected on drug enzyme induction or inhibition such as barbitals within 30 days prior to study medication dosing
* Subjects who have continuously consumed grapefruit juice or caffeine (grapefruit juice or caffeine > 5 cups/day), or who can't refrain from intake during hospitalization
* Subjects who have continued to drink alcohol (alcohol> 30 g/day) or who can't quit drinking during hospitalization
* Severe heavy smoker(cigarette > 10 cigarettes per day) or subjects who can't quit smoking during hospitalization
* Subjects that the investigator deems unsuitable for participation in the clinical trial due to laboratory test results or other excuse such as non-responding to request or instruction by investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-22 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration at steady state(Cmax,ss) of HL237 | 0(before dosing), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hour(after dosing) on day 21 and day 22
  Comparison of pharmacokinetic parameters between when administered tacrolimus with HL237 and without HL237
Area under the plasma concentration versus time curve during a dosage interval(AUCτ) of HL237 | 0(before dosing), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hour(after dosing) on day 21 and day 22
  Comparison of pharmacokinetic parameters between when administered tacrolimus with HL237 and without HL237
Peak whole-blood concentration(Cmax) of tacrolimus | 0(before dosing), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72hour(after dosing) on day 1 and day 22
  Comparison of pharmacokinetic parameters between when administered tacrolimus with HL237 and without HL237
Area under the whole-blood concentration versus time curve from time zero to time of last measurable concentration(AUClast) of tacrolimus | 0(before dosing), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72hour(after dosing) on day 1 and day 22
  Comparison of pharmacokinetic parameters between when administered tacrolimus with HL237 and without HL237

CONTACTS AND LOCATIONS:
Locations (1):
- The Korea Univertisy Anam Hospital, Seoul, South Korea